CLINICAL TRIAL: NCT07029867
Title: Efficacy and Safety of Traditional Chinese Mecicine Yishen Daluo Yin Granule for Relapsing-remitting Multiple Sclerosis: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Yishen Daluo Yin Granule for Relapsing-Remitting Multiple Sclerosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ying Gao (Other)
Collaborators: First Affiliated Hospital of Jinan University (Other); The Second Hospital of Hebei Medical University (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor-Investigator, Ying Gao, Professor, Dongzhimen Hospital, Beijing
Organization: Dongzhimen Hospital, Beijing (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024DZMEC-604
Record Dates: First submitted 2025-06-09; First posted 2025-06-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-05

CONDITIONS: Relapse Remitting Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YSDLY group (Experimental): RRMS patients received YSDLY granuls.
  Interventions: Drug: Yishen Daluo Yin granuls
- Placebo group (Placebo Comparator): RRMS patients received placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Yishen Daluo Yin granuls — The patient takes YSDLY granules or placebo twice a day.
  Arms: YSDLY group
Drug: Placebo — The patient takes placebo (YSDL mimetic granules) twice a day.
  Arms: Placebo group

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of YSDLY granule in patients with RRMS. This will be a multi-center, randomized, double-blind, placebo-controlled study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 to 55 when signing the informed consent, with no gender restrictions.
2. Participants meet the diagnostic criteria for multiple sclerosis (MS) as outlined in the 2017 McDonald's diagnostic criteria and the 2023 edition of the Chinese Guidelines for the Diagnosis and Treatment of Multiple Sclerosis.
3. No clinical relapse, as defined in the protocol, has occurred for 30 days or more prior to screening and baseline (Day 1), and neurological function remains stable.
4. At least 1 relapse with evidence within two years prior to screening is required. This can be demonstrated by: a. Evidence of one relapse within one year prior to screening; b. At least one gadolinium-enhanced T1 lesion on MRI within the six months prior to screening.
5. Participants with EDSS scores ranging from 0 to 5.5 at screening and baseline (Day 1) are eligible for inclusion. However, patients with an EDSS score of ≤ 2 at screening may only be included if their disease duration does not exceed 10 years.
6. Women who were tested for fertility had negative results for pregnancy in their urine during the screening period, prior to the first day of medication.
7. Signing the informed consent form, which the participant must fully understand, indicates that the individual has been provided with all pertinent information regarding the trial prior to enrollment and agrees to adhere to the protocol's requirements.

Exclusion Criteria:

1. According to the 2017 McDonald's guidelines and the 2023 version of the Chinese Multiple Sclerosis Diagnosis and Treatment Guidelines, individuals diagnosed with progressive MS, including both primary progressive MS (PPMS) and secondary progressive MS (SPMS), are excluded.
2. Participants with an EDSS score of 2.0 or lower and a disease duration of more than 10 years during the screening process.
3. Participants diagnosed with an immune system disease other than MS, or any other condition requiring oral, intravenous, or intramuscular corticosteroid medications, except for well-controlled type 2 diabetes or thyroid disease.
4. Active and clinically significant viral, bacterial, tuberculosis, or fungal infections, as well as any severe acute infection that requires hospitalization or treatment with parenteral antibiotics within four weeks prior to screening; participants who have had close contact with patients suffering from infectious diseases, such as active tuberculosis; individuals who have tested positive for human immunodeficiency virus (HIV) either in the past or during screening; and those who have tested positive for hepatitis C virus (HCV) RNA or have a hepatitis B virus (HBV) DNA level of ≥ 10^6 copies/mL in the past or during screening.
5. Participants with a history of any serious or life-threatening bleeding events, such as hemophilia, other coagulation disorders, or an international normalized ratio (INR) of 1.5 or greater, or an activated partial thromboplastin time (APTT) of 1.5 times the upper limit of the laboratory reference range (ULN), are excluded.
6. Participants who have experienced an acute myocardial infarction or cerebrovascular disease within six months after screening, currently have active angina, or have a history of congestive heart failure that meets New York Heart Association (NYHA) Class III or IV criteria are excluded. Additionally, participants with long-term uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg), those with electrocardiogram (ECG) abnormalities or any other significant active medical conditions that the researchers believe may affect their participation are also excluded.
7. There are other clinically significant abnormalities that researchers deem important, as well as major surgical procedures conducted within the two months preceding the screening.
8. Participants have experienced episodes of severe depression within the six months prior to the screening, or are unable to complete this study due to mental illness, cognitive disorders, or emotional disorders.
9. Participants with a history of cancer (unless cured>5 years), or any other illness with a life expectancy of less than 1 year.
10. Pregnant or lactating women, or women of childbearing age who have a negative pregnancy test during screening but refuse to take effective contraceptive measures.
11. Participants with an estimated glomerular filtration rate (eGFR) of less than 30 mL/min/1.73 m², or those with any kidney disease that contraindicates the use of gadolinium, such as acute kidney injury. The formula for calculating eGFR is: eGFR = 186 × (blood creatinine)-¹.⁵⁴ × (age)-⁰.²⁰³ × (0.742 if female). The unit for blood creatinine is mg/dL, and the unit for age is years.
12. ALT and AST levels greater than 2 times the upper limit of normal (ULN), total bilirubin levels exceeding 1.5 times the ULN, or any other clinically significant laboratory abnormalities.
13. Significant reductions in blood cell counts, including a neutrophil count of less than 1,500/mm³, a platelet count of less than 75,000/mm³, an absolute lymphocyte count of less than 1,000/mm³, or a white blood cell count of less than 3,500/mm³.
14. Participants who cannot performe MRI scans in certain situations include those with known allergic reactions to gadolinium contrast agents, individuals with pacemakers, or those with other contraindications.
15. Individuals who are suspected or known to be allergic to the investigational drug or its ingredients should be excluded.
16. Participants who have used any of the following medications in the four weeks prior to randomization are excluded: injections (including intravenous or intramuscular), oral corticosteroids, adrenocorticotropic hormone (ACTH), intravenous immunoglobulin, plasma exchange, immunoadsorption therapy, beta interferon, glatiramer acetate, or other fumarate esters such as diimidazole fumarate and dimethyl fumarate, as well as teriflunomide.
17. Individuals who have previously used natalizumab or S1P receptor modulators (such as Fingolimod, Sinimod, Ozamod, etc.) in 12 weeks before randomization.
18. Participants who have used any of the following pharmaceuticals or therapies within 48 weeks prior to randomization are excluded: dalizumab, BTK inhibitors, mitoxantrone, or lymphocyte depletion therapies (such as alemtuzumab, rituximab, ofatumumab, orelizumab, anti-CD4 preparations, cladribine, cyclophosphamide, azathioprine, systemic radiotherapy, bone marrow transplantation, or other therapies not explicitly listed).
19. Dalfampridine or Fampridine can be used as adjuvant therapy if administered at stable doses in 12 weeks prior to randomization.
20. Participants who have have participated in clinical trials of other investigational drugs within the past 48 weeks.
21. Any situation that other researchers deem inappropriate for participation in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients without combined unique active lesions (CUALs) in 24W compared to baseline. | From enrollment to the end of treatment at 24 weeks.
  The proportion of patients without combined unique active lesions (CUALs) at 24 weeks compared to baseline. CUALs refer to newly identified gadolinium-enhanced T1 lesions or newly added or expanded T2 lesions that are not counted repeatedly.

SECONDARY OUTCOMES:
Average Relapse Time | From enrollment to the end of treatment at 24 weeks.
Annual Relapse Rate | From enrollment to week 12 and 24.
Proportion of Patients Without Relapse | From enrollment to week 12 and 24.
Changes in Expanded Disability Status Scale (EDSS) Compared to Baseline. A score of 0 on the scale indicates the absence of clinical symptoms, while a score of 10 represents death resulting from illness. | From enrollment to week 12 and 24.
Number of newly added gadolinium enhanced T1 lesions compared to baseline. | From enrollment to week 12 and 24.
Number of newly added or expanded T2 lesions compared to baseline. | From enrollment to week 12 and 24.
Changes in T2 lesion volume compared with baseline | From enrollment to week 12 and 24.

OTHER OUTCOMES:
Changes in the level of neurofilament light chain (NFL) compared to the baseline | From enrollment to week 12 and 24.
Changes in the multiple sclerosis quality of life questionnaire (MSQol-54) scale scores compared to the baseline. The MSQOL-54 scale has a total score range of 0 to 100 points, with higher scores indicating a better quality of life. | From enrollment to the end of the treatment at 24 weeks.
Changes in the EuroQol Five Dimensions (EuroQol-5D) scale scores compared to the baseline. The higher the score, the better the quality of life. | From enrollment to the end of treatment at 24 weeks.
Changes in TCM syndrome compared to baseline. | From enrollment to week 4, 8, 12, 16, 20, and 24.